CLINICAL TRIAL: NCT03128151
Title: PORCzero: PostOperative Residual Curarization
Brief Title: Reducing the Incidence of PostOperative Residual Curarization
Acronym: PORCzero
Status: Completed | Type: Observational
Sponsor: Oscar Diaz-Cambronero (Other)
Collaborators: Instituto de Investigacion Sanitaria La Fe (Other); Instituto de Investigacion Sanitaria INCLIVA (Other)
Responsible Party: Sponsor-Investigator, Oscar Diaz-Cambronero, Physician, specialist in Anesthesiology, Hospital Universitario La Fe
Organization: Hospital Universitario La Fe (Other)
Other Study IDs: CEO-SUG-2016-01
Record Dates: First submitted 2017-04-10; First posted 2017-04-25 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Neuromuscular Blockade
Keywords: NMB (Neuromuscular Blockade); Anesthesia; Curarization; TOFr (train of four); PACU (postanesthesia care unit); Monitorization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Intraoperative neuromuscular monitoring and pharmacological reversion according to data sheet
  Interventions: Behavioral: Educational program for clinicians: implementation of a package of clinical prevention measures of NMB
- Control group: Treated according to usual clinical practice

INTERVENTIONS:
Behavioral: Educational program for clinicians: implementation of a package of clinical prevention measures of NMB — Intraoperative neuromuscular monitoring and pharmacological reversion of NMB according to data sheet
  Groups: Study group

SUMMARY:
The NMB (Neuromuscular Blockade) is the most frequent complication in anesthesiology associated with an increase in adverse respiratory events in the postoperative period. Its appearance depends on multiple factors. The introduction of a comprehensive educational strategy aimed at promoting the proper management of NMB in the intraoperative period and a package of measures that must be performed (intraoperative neuromuscular monitoring and reversal of the effect of neuromuscular blockers) may contribute to a decrease in the incidence of NMB, Increase safety in the surgical patient and decrease associated costs.

DETAILED DESCRIPTION:
Multicenter, epidemiological, prospective, randomized, sequential study. The introduction of an educational program and a package of clinical measures (specific monitoring and pharmacological reversion) in the incidence of NMB will be evaluated by evaluating variations in this incidence of NMB, the rate of compliance with the preventive measures and the perception of the Safety in the perioperative, through pre and postoperative survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Classification of the American Society of Anesthesiologists (ASA I-III).
* Patients with absence of cognitive deficit.
* Informed informed consent prior to surgery

Exclusion Criteria:

* Negative of the patient to participate in the study
* Patients under the age of 18 or incapable of giving their consent
* ASA IV-V
* Pregnancy or breastfeeding
* Associated neuromuscular disorders
* Diabetes mellitus with diagnosed neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to general anesthesia with neuromuscular blockade, extubated before admission to the Post Anesthesia Recovery Unit
Sampling Method: Probability Sample
Enrollment: 2314 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of PORC. | Six months, first three months to evaluate PORC incidence and then three months to evaluate PORC incidence after educational intervention.
  To reduce the incidence of PORC ≤ 10% by the introduction of an educational program and a bundle of preventive measures (including intraoperative monitoring and reversal of neuromuscular blocking agents (NMBA)).

SECONDARY OUTCOMES:
Compliance rate with the bundle of measures | Six months, first three months to evaluate PORC incidence and then three months to evaluate PORC incidence after educational intervention.
  To evaluate if the educational program increases compliance of clinical preventive measures, if the reduction of incidence of BNMR is maintained, and, in addition, if this compliance is maintained over time.
Rate of intraoperative monitoring | Six months, from the beginning, with no intervention, until the end of phase III (end of recruitment in both groups).
  Rate of compliance of clinical prevention measures with intraoperative monitoring.
Rate of reversal of NMBA | Six months, from the beginning, with no intervention, until the end of phase III (end of recruitment in both groups).
  Rate of compliance of clinical prevention measures with NMBA reversal after surgery.
Perception of safety -increase- by anesthesiologists | Six months, from the beginning, with no intervention, until the end of phase III (end of recruitment in both groups).
  To evaluate, from the point of view of patient safety, whether the perception of safety by clinicians is maintained, through a survey before and after the intervention.
Incidence of postoperative adverse events. | Six months, from the beginning, with no intervention, until the end of phase III (end of recruitment in both groups).
  Incidence of postoperative complications in relation to the NMB reversal rate.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Diaz Cambronero, MD, Principal Investigator — Hospital La Fe
Locations (1):
- Hospital la Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Diaz-Cambronero O, Mazzinari G, Errando CL, Garutti I, Gurumeta AA, Serrano AB, Esteve N, Montanes MV, Neto AS, Hollmann MW, Schultz MJ, Argente Navarro MP; Reducing the Incidence of Post Operative Residual Curarization Zero investigators. An educational intervention to reduce the incidence of postoperative residual curarisation: a cluster randomised crossover trial in patients undergoing general anaesthesia. Br J Anaesth. 2023 Sep;131(3):482-490. doi: 10.1016/j.bja.2023.02.031. Epub 2023 Apr 20. PMID 37087332